CLINICAL TRIAL: NCT01637558
Title: Optimal Dosing of 1st Line Antituberculosis and Antiretroviral Drugs in Children (a Pharmacokinetic Study)
Acronym: DATiC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Liverpool School of Tropical Medicine (Other); Uppsala University (Other); University of North Carolina (Other)
Responsible Party: Principal Investigator, Helen Margaret McIlleron, Assistant Prof, University of Cape Town
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DATiC
Record Dates: First submitted 2012-07-02; First posted 2012-07-11 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Tuberculosis; HIV
MeSH Terms: conditions — Tuberculosis | interventions — Nevirapine; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Main TB cohort (No Intervention): Children with tuberculosis 0-12 years of age
- Lopinavir/Ritonavir - Cases (Experimental): children 3-20 kg with tuberculosis and indication for LPV/r-based ART
  Interventions: Drug: 8 hourly LPV/r during TB treatment
- Lopinavir/Ritonavir - Controls (Experimental): Children 3-20 kg on LPV/r-based ART; no TB
  Interventions: Drug: Lopinavir/Ritonavir
- Nevirapine arm (Experimental): children with TB and indication for nevi rapine-based ART
  Interventions: Drug: Nevirapine

INTERVENTIONS:
Drug: 8 hourly LPV/r during TB treatment — 8 hourly LPV/r during TB treatment
  Arms: Lopinavir/Ritonavir - Cases
Drug: Nevirapine
  Arms: Nevirapine arm
Drug: Lopinavir/Ritonavir
  Arms: Lopinavir/Ritonavir - Controls

SUMMARY:
The aims of this project are to:

1. To evaluate the pharmacokinetics of first line antituberculosis drugs (isoniazid, rifampicin, pyrazinamide and ethambutol) when applying the 2010 WHO/IUATLD dosing guidelines across pediatric populations (0-12 years of age, HIV infected and uninfected, and with varied nutritional status) in Cape Town, South Africa and Blantyre, Malawi.
2. To evaluate an 8-hourly weight band-based dosing strategy for lopinavir/ritonavir using the commercially available lopinavir/ritonavir (4:1 ratio) in children in South Africa receiving rifampicin-based antituberculosis treatment.
3. To evaluate the pharmacokinetics of nevirapine in children in Malawi receiving rifampicin-based antituberculosis treatment.

DETAILED DESCRIPTION:
HIV and tuberculosis are a major public health problem in children. Challenges to treat children with tuberculosis include a lack of knowledge about optimal dosing of first line antituberculosis drugs across ages, nutritional status and HIV infection status, the absence of an appropriate regimen to co-administer rifampin and lopinavir/ritonavir, the key first line drugs for tuberculosis and HIV, and uncertainty about NVP exposure in young children during rifampin-based tuberculosis therapy.

In total, 240 children < 12 years of age with tuberculosis will be enrolled at Red Cross Children's Hospital in Cape Town and Queen Elizabeth Central Hospital, Blantyre. In the second month of antituberculosis treatment, one dose of the drugs in their first-line regimens will be administered according to 2010 WHO/IUATLD guidelines (study drugs) and blood will be sampled for pharmacokinetic analysis over the following 8-10 hours.

Children on antiretroviral treatment (started prior to or during TB treatment) will receive 2 weeks of antiretrovirals (lopinavir/ritonavir or nevirapine) according in the study doses (adjusted 8 hourly doses of lopinavir/ritonavir, or nevirapine doses according to WHO's recommended weight band-based doses) in combination with antituberculosis treatment, prior to pharmacokinetic assessments of both antiretroviral and antituberculosis drugs. Children receiving nevirapine will also undergo pharmacokinetic evaluation 1 month after completion of antituberculosis treatment to evaluate nevirapine concentrations in the absence of antituberculosis drugs. In addition to the 240 children with tuberculosis, 25 HIV infected South African children without tuberculosis will be recruited to evaluate lopinavir concentrations in the absence of antituberculosis drugs.

A population approach will be used to estimate the optimal doses of rifampicin, isoniazid, pyrazinamide and ethambutol in children according to covariates (e.g. age, weight, HIV status, nutritional status) found to have an important influence on the drug concentrations. Similarly population models will be used to describe lopinavir/ritonavir and nevirapine pharmacokinetics in children receiving rifampicin-based antituberculosis treatment, evaluate the dosing approaches and to simulate alternative optimal dosing approaches as indicated.

ELIGIBILITY:
Inclusion Criteria:

ALL STUDY PARTICIPANTS

* Aged < 12 years.
* Weighing > 1.5 kg and < 30 kg.
* Written informed permission of parent or legal guardian for their child to participate.
* Absence of clear indication of unwillingness or refusal to participate, and in children > 7 years of age, assent to participate.
* No contraindications to PK sampling (children with obviously very poor venous access will not be included).
* Able to comply with study visits and procedures including regular adherence to routine medication, and adherence to the study medication.
* Enrollment will be deferred in children with acute severe illness which would likely jeopardize participation (such as illness causing severe respiratory impairment, acute severe diarrhea, acute central nervous system impairment, severe life threatening systemic illness, or other severe conditions requiring hospitalization which would jeopardize participation). Children may be enrolled after recovery from acute illness.

ADDITIONAL CRITERIA FOR THE MAIN TB COHORT AND SUBSTUDIES

1. Main TB cohort

   INCLUSION A recent diagnosis of TB and receiving intensive phase antiTB treatment with 1st-line drugs (rifampicin, isoniazid, pyrazinamide with or without ethambutol, in standard doses).
2. LPV SUBSTUDY

   CASES & CONTROLS
   * Children in whom ART with a LPV/r-containing regimen is indicated, OR, Children established on a LPV/r-containing regimen.
   * ALT < 5-times the upper limit of the normal range.
   * Children weighing 3.0 - 19.9 kg.
   * Neonates must have a postmenstrual age of at least 42 weeks and a postnatal age of at least 14 days.

   CASES

   - HIV infected children enrolled to the main cohort with at least 2 weeks remaining before the end of intensive phase antiTB treatment such that PK sampling can be scheduled after 2 weeks of combined ART and antiTB treatment, but before the continuation phase of antiTB treatment is started.

   CONTROLS

   - HIV infected children without TB.

   Weighted enrollment of controls will be performed such that the number of controls in each of the age groups < 6 months, 6 months to 2 years, and > 2 years, will be approximately equal to the numbers of cases in those age groups. As most of the children with TB will be started on ART after their TB diagnosis, recruitment of controls will be focused on children who have recently started ART (on treatment < 3 months).
3. NVP SUBSTUDY

   * HIV infected children receiving intensive phase antiTB treatment and enrolled to the main study cohort
   * Started on ART including NVP (in WHO's recommended weight band-based doses) and 2 nucleoside reverse transcriptase inhibitors.

Exclusion Criteria:

* Indication for increased or reduced doses of 1st-line antiTB drugs (e.g. marked hepatic or renal impairment, TB meningitis).

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve (AUC) for rifampicin, isoniazid, pyrazinamide, ethambutol, lopinavir and nevirapine | 5 years
  Population PK model-derived AUC's (in mg.h/L)for each of the first line anti-TB drugs, and for the substudies, lopinavir and nevirapine respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Helen M McIlleron, PhD, Principal Investigator — University of Cape Town; Heather Zar, PhD, Principal Investigator — University of Cape Town
Locations (4):
- Queen Elizabeth Central Hospital, Blantyre, Malawi
- South Africa (3):
  - Red Cross Childrens Hospital, Cape Town, Western Cape
  - KIDCRU, Tygerberg Hospital, Department of Paediatrics and Child Health, Stellenbosch University, South Africa., Cape Town, Western Cape
  - Desmond Tutu Centre, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Galileya LT, Wasmann RE, Chabala C, Rabie H, Lee J, Njahira Mukui I, Hesseling A, Zar H, Aarnoutse R, Turkova A, Gibb D, Cotton MF, McIlleron H, Denti P. Evaluating pediatric tuberculosis dosing guidelines: A model-based individual data pooled analysis. PLoS Med. 2023 Nov 21;20(11):e1004303. doi: 10.1371/journal.pmed.1004303. eCollection 2023 Nov. PMID 37988391
- [Derived] Rabie H, Rawizza H, Zuidewind P, Winckler J, Zar H, Van Rie A, Wiesner L, McIlleron H. Pharmacokinetics of adjusted-dose 8-hourly lopinavir/ritonavir in HIV-infected children co-treated with rifampicin. J Antimicrob Chemother. 2019 Aug 1;74(8):2347-2351. doi: 10.1093/jac/dkz171. PMID 31081020
- [Derived] Bekker A, Schaaf HS, Draper HR, van der Laan L, Murray S, Wiesner L, Donald PR, McIlleron HM, Hesseling AC. Pharmacokinetics of Rifampin, Isoniazid, Pyrazinamide, and Ethambutol in Infants Dosed According to Revised WHO-Recommended Treatment Guidelines. Antimicrob Agents Chemother. 2016 Mar 25;60(4):2171-9. doi: 10.1128/AAC.02600-15. Print 2016 Apr. PMID 26810651